CLINICAL TRIAL: NCT06812858
Title: A Multicenter Prospective Phase II Study Evaluating the Efficacy and Safety of PD-1 Inhibitors Maintenance in Patients With Refractory/Relapsed Classical Hodgkin Lymphoma After Autologous Hematopoietic Stem Cell Transplantation
Brief Title: PD-1 Inhibitors Maintenance for cHL Post-autoHCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29/24-н
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Classic Hodgkin lymphoma; autologous hematopoietic stem cell transplantation; nivolumab; pembrolizumab
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 Inhibitors maintenance (Experimental)
  Interventions: Drug: Nivolumab, Pembrolizumab

INTERVENTIONS:
Drug: Nivolumab, Pembrolizumab — The choice of drug and its dose for maintenance therapy is at the discretion of the study centre (e.g. nivolumab, pembrolizumab). Maintenance therapy should be initiated no later than 60 days after D0, exceptions may be made due to reasonable justification in consultation with the Study PI and will not be considered a protocol deviation.
  Nivolumab maintenance therapy regimens:
  * Nivolumab (40 mg, fixed dose) IV D1 of each 14-days cycle up to 12 cycles
  * Nivolumab (3 mg/kg) IV D1 of each 14-days cycle up to 12 cycles
  Pembrolizumab maintenance therapy regimen:
  -Pembrolizumab (200 mg, fixed dose) IV D1 of each 21-days cycle up to 8 cycles

SUMMARY:
This phase II study is designed to determine the clinical efficacy of PD-1 inhibitors, administered as maintenance therapy after autologous stem cell transplant (autoHCT), in patients with relapsed or refractory (R/R) classical Hodgkin Lymphoma (cHL)

DETAILED DESCRIPTION:
Classic Hodgkin lymphoma (cHL) accounts for about 10-30% of all malignant lymphomas and predominantly occurs in individuals of working age. Thanks to modern chemoradiotherapy methods, a durable remission is achieved in 80% of patients. However, for a significant proportion of patients, achieving a sustained remission after first-line chemotherapy is not possible. The standard treatment for patients with refractory/relapsed cHL is second-line intensified chemotherapy followed by high-dose chemotherapy with autologous hematopoietic stem cell transplantation (auto-HSCT). While this approach allows some patients to achieve long-lasting remission, more than 50% of them experience disease progression or relapse. Current therapeutic strategies for such patients are limited and often fail to produce long-term remission. Given that most relapses occur within the first two years after auto-HSCT, a maintenance therapy strategy aimed at preventing relapse and disease progression is a promising avenue for improving outcomes in this patient group.

In 2015, based on the results of the AETHERA study, the U.S. Food and Drug Administration (FDA) approved the use of brentuximab vedotin (BV) as consolidation therapy for patients with cHL at high risk of relapse or progression following auto-HSCT. BV demonstrated an increase in median progression-free survival (PFS), with 42.9 months in the BV group compared to 24.1 months in the placebo group. However, despite this improvement, the two-year PFS among patients receiving BV was only 63%. Moreover, in the AETHERA study, with a planned 16 cycles of BV therapy, 23% of patients discontinued maintenance therapy due to severe adverse events, and 31% required dose reductions because of peripheral neuropathy.

Currently, there are data from several studies on the safety and efficacy of PD-1 inhibitor maintenance therapy for patients with cHL. In a small phase II trial, 30 patients (90% with high-risk factors) received up to 8 cycles of pembrolizumab (200 mg every 3 weeks) as maintenance therapy after auto-HSCT. The 18-month PFS rate was 82%, with an overall survival (OS) of 100% (Armand et al.). Similar results were obtained with nivolumab (240 mg every 3 weeks) as maintenance therapy. Preliminary findings showed a 6-month PFS of 92% and OS of 100%. These studies also demonstrated an acceptable toxicity profile: therapy discontinuation due to adverse events occurred in 17% of patients receiving pembrolizumab and in 10% of those on nivolumab maintenance therapy.

Data have also been obtained on the efficacy of a fixed-dose nivolumab regimen (40 mg every 2 weeks) for patients with r/r cHL: the objective response rate was 70%, and the 18-month PFS was 53.6%. Based on these results, the fixed-dose 40 mg nivolumab regimen, which showed comparable efficacy for this patient group, has been included in the draft Russian clinical guidelines for the diagnosis and treatment of patients with r/r cHL.

Thus, the use of PD-1 inhibitors, having a favorable toxicity profile, may achieve durable remissions in patients with cHL after auto-HSCT. Moreover, the available data indicating comparable efficacy of a fixed-dose nivolumab regimen versus the standard approach increases the accessibility of this treatment option. Employing PD-1 inhibitors is an important step in modifying the therapy strategy for patients with r/r cHL and in preventing relapses in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years;
* Diagnosis of r/r cHL with auto-HCT being performed as consolidation of 2 or later therapy lines;
* High-risk cHL (Primary refractoriness after first-line therapy / Relapse after first line therapy within 12 months / PET/CT-positive status at the time of auto-HCT / Late relapse (> 12 months) with unfavourable prognosis factors (extranodal lesion and/or bulky and/or B-symptoms) / More than one salvage regimen performed)
* Complete or partial response by PET/CT after auto-HSCT
* No evidence of grade 3-4 adverse events (CTCAEs) after auto-HCT at the time of inclusion in the study;
* Achieved recovery of peripheral blood counts after auto-HSCT (white blood cell count> 1 109/L, absolute neutrophil count> 0.5 109/L, platelets > 25 109/L);
* ECOG 0-2; The decision to include patients that do not fulfil the criteria of hight-risk cHL is made in consultation with the PI

Exclusion Criteria:

* Patients who have received PD1-inhibitor therapy in the previous lines of treatment and had to interrupt treatment early due to the development of adverse events of therapy;
* Severe organ failure: creatinine values more than 2 ULN; ALT, AST more than 5 ULN; bilirubin more than 1.5 ULN;
* Respiratory failure of more than 1 degree at the time of inclusion in the study;
* Unstable haemodynamics at the time of inclusion in the study;
* Acute bacterial, viral or fungal infection at the time of inclusion;
* Active autoimmune diseases (subjects with type 1 diabetes mellitus and hypothyroidism requiring only hormone replacement therapy, and skin diseases such as vitiligo, allopecia, or psoriasis that do not require systemic therapy may be eligible);
* Pregnancy or breastfeeding, or planning pregnancy or parenthood during the study period;
* Somatic or psychiatric pathology that prevents the signing of informed consent;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of PD-1 inhibitors as maintenance therapy after autoHCT in patients with r/r cHL, as assessed by 24-month progression-free surviva | From the first dose of study treatment to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed at 24 months

SECONDARY OUTCOMES:
To determine the 12- and 18-month PFS in patients with r/r cHL receiving PD-1 inhibitors as maintenance therapy following auto-HSCT. | From the first dose of study treatment to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed at 12 or 18 months
To determine the 12-, 18-, and 24-month overall survival (OS) in patients with r/r cHL receiving PD-1 inhibitors as maintenance therapy following auto-HSCT. | From the first dose of study treatment to death from any cause, assessed up to 12, 18 and 24 months
To determine the 12-, 18-, and 24-month cumulative incidence of relapse (CIR) in patients with r/r cHL receiving PD-1 inhibitors as maintenance therapy following auto-HSCT. | Up to 12, 18 and 24 months
To establish the safety and tolerability of PD-1 inhibitors in the maintenance setting, defined as the frequency, severity, and spectrum of adverse events (AEs) | observed during therapy and for one year following completion of maintenance therapy.
  Incidence of toxicities evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Mikhailova, MD, Study Chair — St. Petersburg State Pavlov Medical University
Locations (3):
- National Research Oncology Center, Astana, Kazakhstan
- Russia (2):
  - National Medical and Surgical Center named after N.I. Pirogov, Moscow
  - RM Gorbacheva Research Institute, Pavlov University, Saint Petersburg